CLINICAL TRIAL: NCT00808808
Title: Assessing Choice in the Employer Setting (ACES Study): An Observational Study to Assess the Impact of Offering Intranasal Vaccine on Influenza Vaccination Rates in the Employer Setting
Brief Title: Assessing Choice in the Employer Setting (ACES) Study
Acronym: MA181
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Collaborators: Passport Health (Industry); University of Pittsburgh (Other)
Responsible Party: Seth Toback, MD, Medimmune LLC
Other Study IDs: MI-MA-181
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: FluMist, TIV, vaccination rates
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm A (Control): A control arm of usual care offering TIV with baseline advertisement
  Interventions: Biological: Control - Usual care offering TIV only with baseline advertisement
- Arm B (Choice): An intervention arm offering choice of TIV or FluMist with baseline advertisement, including advertisement to highlight the availability of FluMist
  Interventions: Biological: Choice of TIV or FluMist with baseline advertisement
- Arm C (Choice Plus): An intervention arm offering choice of TIV or FluMist with enhanced advertisement and additional incentives for receiving an influenza vaccination
  Interventions: Other: Choice of TIV or FluMist with enhanced advertisement and incentives

INTERVENTIONS:
Biological: Choice of TIV or FluMist with baseline advertisement — An intervention arm offering choice of TIV or FluMist with baseline advertisement, including advertisement to highlight the availability of FluMist
  Groups: Arm B (Choice)
Other: Choice of TIV or FluMist with enhanced advertisement and incentives — An intervention arm offering choice of TIV or FluMist with enhanced advertisement and additional incentives for receiving an influenza vaccination
  Groups: Arm C (Choice Plus)
Biological: Control - Usual care offering TIV only with baseline advertisement — A control arm of usual care offering TIV with baseline advertisement
  Groups: Arm A (Control)

SUMMARY:
The purpose of this study is to determine, among adults and in the total population, the effects of offering a choice of FluMist or trivalent inactivated vaccine (TIV) in the employer setting when compared to a control group.

DETAILED DESCRIPTION:
The primary objective is to determine, among adults in the 18-49 year old population and in the total population, the effects of offering a choice of FluMist or TIV with and without enhanced advertisement/added incentive on the overall influenza vaccination rates in the employer setting when compared to a control group.

ELIGIBILITY:
Inclusion Criteria for employer sites:

* Located in the United States
* Has not previously offered FluMist in an employee vaccination program in the past or FluMist represented less than 5% of all vaccine received at past programs
* Data are available that will allow for a reliable estimate of the employee (total and 18-49 year old populations) vaccination rate for the 2007-2008 influenza season

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults at least 18 years of age who are current employees attending the influenza clinic sponsored by their employer
Sampling Method: Non-Probability Sample
Enrollment: 4411 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Toback, M.D., Study Director — MedImmune LLC
Locations (37):
- United States (37):
  - Chatsworth, California
  - Novato, California
  - Sacramento, California
  - San Francisco, California
  - Santa Clara, California
  - Santa Monica, California
  - Sunnyvale, California
  - Thousand Oaks, California
  - Boulder, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Hebron, Kentucky
  - La Grange, Kentucky
  - Lawrenceburg, Kentucky
  - Louisville, Kentucky
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Calverton, Maryland
  - Cockeysville, Maryland
  - Columbia, Maryland
  - Crofton, Maryland
  - Hanover, Maryland
  - Hunt Valley, Maryland
  - Laurel, Maryland
  - Sparks, Maryland
  - Basking Ridge, New Jersey
  - Larwenceville, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Rochester, New York
  - High Point, North Carolina
  - Cincinnati, Ohio
  - Hamilton, Ohio
  - Lebanon, Ohio
  - West Chester, Ohio
  - Fredericksburg, Virginia

REFERENCES:
- [Result] Lin CJ, Nowalk MP, Toback SL, Rousculp MD, Raymund M, Ambrose CS, Zimmerman RK. Importance of vaccination habit and vaccine choice on influenza vaccination among healthy working adults. Vaccine. 2010 Nov 10;28(48):7706-12. doi: 10.1016/j.vaccine.2010.07.009. Epub 2010 Jul 16. PMID 20638452
- [Result] Nowalk MP, Lin CJ, Toback SL, Rousculp MD, Eby C, Raymund M, Zimmerman RK. Improving influenza vaccination rates in the workplace: a randomized trial. Am J Prev Med. 2010 Mar;38(3):237-46. doi: 10.1016/j.amepre.2009.11.011. Epub 2009 Dec 24. PMID 20036102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential employers estimated to have at least 60 employees were contacted to determine their interest in participating in the study and were offered an influenza vaccine clinic on site at no cost. A screening questionnaire to determine eligibility was completed. Sites were excluded according to the study inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Started | 4078 (Started includes all employees at participating sites.) | 3757 (Started includes all employees at participating sites) | 4387 (Started includes all employees at participating sites.)
Vaccinated | 1392 (Vaccinated includes all employees who were vaccinated at the employee vaccination clinics.) | 1489 (Vaccinated includes all employees who were vaccinated at the employee vaccination clinics.) | 2132 (Vaccinated includes all employees who were vaccinated at the employee vaccination clinics.)
Completed | 1261 (Completed includes vaccinated employees who completed surveys.) | 1320 (Completed includes vaccinated employees who completed surveys.) | 1830 (Completed includes vaccinated employees who completed surveys.)
Not Completed | 2817 | 2437 | 2557
Not completed — Vaccinated; survey not completed | 131 | 169 | 302
Not completed — Employee was not vaccinated. | 2686 | 2268 | 2255

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus) | Total
Number analyzed (Participants) | 1392 | 1489 | 2132 | 5013
Age, Customized [Number; unit: participants]
  18 to 49 years | 983 | 988 | 1398 | 3369
  ≥ 50 years | 409 | 501 | 734 | 1644
Sex/Gender, Customized [Number; unit: participants] — Includes all vaccinated employees, not only participants who completed surveys.
  participants
    Male | 748 | 814 | 808 | 2370
    Female | 644 | 675 | 1324 | 2643

OUTCOME MEASURES:

1. Primary Outcome: Overall Vaccination Rate, All Ages
Time Frame: 30Sep2008 through 23Dec2008
Population: All employees at participating sites, including those who were vaccinated and those who were not
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Number analyzed (Participants) | 4078 | 3757 | 4387
Percentage of participants | 41.6 | 45.1 | 51.0

2. Primary Outcome: Overall Vaccination Rate, Employees 18 to 49 Years of Age
Time Frame: 30Sep2008 through 23Dec2008
Population: All vaccinated employees at participating sites, including those who completed surveys and those who did not
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Number analyzed (Participants) | 983 | 988 | 1398
Percentage of participants | 38.5 | 40.9 | 46.1

3. Secondary Outcome: Change in Influenza Vaccination Rate From Baseline Season to Intervention Season in the Total Population
Description: Rate difference by arm from baseline to intervention season
Time Frame: 2007-2008 season through 2008-2009 season
Population: All vaccinated employees at participating sites, including those who completed surveys and those who did not
Measure: Number; unit: percentage points
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Number analyzed (Participants) | 1392 | 1489 | 2132
percentage points | 4.7 | 4.8 | 12.7

4. Secondary Outcome: Change in Influenza Vaccination Rate From Baseline Season to Intervention Season in Employees 18-49 Years of Age
Description: Rate difference by arm from baseline to intervention season
Time Frame: 2007-2008 season through 2008-2009 season
Population: All vaccinated employees 18-49 years of age at participating sites, including those who completed surveys and those who did not
Measure: Number; unit: percentage points
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Number analyzed (Participants) | 983 | 988 | 1398
percentage points | 3.7 | 2.4 | 9.7

5. Secondary Outcome: Percent of Eligible Participants 18-49 Years of Age Choosing FluMist During Intervention Season
Time Frame: 30Sep2008 through 23Dec2008
Population: as for outcome 4
Measure: Number; unit: percent
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Number analyzed (Participants) | 983 | 988 | 1398
percent | 0.8 | 19.1 | 26.8

6. Secondary Outcome: Characteristics of Participants 18-49 Years of Age Choosing FluMist vs TIV: Race
Description: Percent of participants 18-49 years of age who chose FluMist vs TIV for influenza vaccination and who self-identified as white
Time Frame: 30Sep2008 through 23Dec2008
Population: All participants who completed surveys and were eligible to receive FluMist
Measure: Number; unit: percent
Groups:
- Vaccinated With FluMist: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with FluMist, and who self-identified as white
- Vaccinated With TIV: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with TIV, and who self-identified as white.
Arm/Group | Vaccinated With FluMist | Vaccinated With TIV
Number analyzed (Participants) | 399 | 1990
percent | 67.8 | 71.8

7. Secondary Outcome: Characteristics of Participants 18-49 Years of Age Choosing FluMist vs TIV: Education
Description: Percent of participants 18-49 years of age who chose FluMist vs TIV for influenza vaccination and who self-identified as college graduates.
Time Frame: 30Sep2008 through 23Dec2008
Population: All participants who completed surveys and were eligible to receive FluMist
Measure: Number; unit: percent
Groups:
- Vaccinated With FluMist: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with FluMist, and who self-identified as college graduates.
- Vaccinated With TIV: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with TIV, and who self-identified as college graduates.
Arm/Group | Vaccinated With FluMist | Vaccinated With TIV
Number analyzed (Participants) | 399 | 1990
percent | 73.4 | 52.8

8. Secondary Outcome: Characteristics of Participants 18-49 Years of Age Choosing FluMist vs TIV: Gender
Description: Percent of participants 18-49 years of age who chose FluMist vs TIV for influenza vaccination and who self-identified as male.
Time Frame: 30Sep2008 through 23Dec2008
Population: All participants who completed surveys and were eligible to receive FluMist
Measure: Number; unit: percent
Groups:
- Vaccinated With FluMist: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with FluMist, and who self-identified as male.
- Vaccinated With TIV: Characteristics of vaccinated employees 18-49 years of age who were eligible for FluMist and chose vaccination with TIV, and who self-identified as male.
Arm/Group | Vaccinated With FluMist | Vaccinated With TIV
Number analyzed (Participants) | 399 | 1990
percent | 49.9 | 49.7

ADVERSE EVENTS:
Time Frame: September 2008 - December 2008
Description: Participants received commercial vaccine per routine care at employer clinics; no investigational treatment was given. Safety data were not collected. Any participant who experienced an adverse event associated with a MedImmune commercial vaccine was to be advised to notify the MedImmune Patient Safety Department. No such events were reported.
Arm/Group | Arm A (Control) | Arm B (Choice) | Arm C (Choice Plus)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was conducted during a single season, data to evaluate effects of the intervention by race were unavailable, baseline vaccination data were available at the company level only, and vaccines received outside the workplace were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.The principal investigators (PIs) also agree for data to be presented first as a joint, multi-center publication.